CLINICAL TRIAL: NCT05729919
Title: Healing Dynamics of Free Gingival Grafts; a Colorimetric and Volumetric Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Principal Investigator Gonzalo Blasi, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2020-08
Record Dates: First submitted 2023-01-13; First posted 2023-02-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Free Gingival Graft
Keywords: FGG; Volume; Color

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Free gingival graft (Experimental): Free gingival technique will be done
  Interventions: Procedure: Free gingival graft technique

INTERVENTIONS:
Procedure: Free gingival graft technique — A horizontal partial thickness incision will be trace at the MGJ to dissect the alveolar mucosa from the keratinized tissue. The alveolar mucosa will be dissected from the underlying periosteum to create an envelope of 4-5 mm apical to the bone dehiscence associated with the gingival recessions. The keratinized tissue coronal to the first incision and neighboring the recession will be de-epithelialized to expose the connective tissue and create a trapezoidal recipient bed having a large apical base at the MGJ and a narrower coronal base just coronal to the CEJ of the experimental units. The grafts will be taken from the palate.The grafts will be positionned with the coronal edge of the CEJ.
  Interrupted sutures (6-0 polypropylene, prolene) will be positionned to stabilize the graft. Sling crossed sutures anchored to the periosteum apical to the graft and placed to ensure a tight adaptation of the graft to the root surface

SUMMARY:
Gingival recession on vestibular surfaces of teeth is a frequent occurrence in patients with high standards of oral hygiene, affecting all types of teeth. During the last three decades, several surgical techniques have been proposed to treat single and multiple gingival recessions: pedicled flaps (laterally displaced (CDL) or coronally advanced (ACC) flaps), free gingival grafts (IGL), bilaminar techniques or procedures regenerative.

DETAILED DESCRIPTION:
One month before surgery, an interview and periodontal therapy (pre-surgical prophylaxis, oral hygiene instructions and brushing technique teaching) will be carried out.

A digital scan of the arch with the teeth to be treated will be made before the surgery, during the surgery (recipient bed and with sutures), at 6 weeks, 3 months, 6 months and 1 year.

On the day of surgery, the recipient bed will be prepared and a free gingival graft will be taken from the palate to cover the exposed root surface or gain keratinized gingiva.

In terms of aesthetics, morbidity and satisfaction will be evaluated through questions.

At 6 weeks, 3 months, 6 months and 1year, the color of the gum will be evaluated using a spectrophotometer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 90 years old
* Patients exhibiting deficient KT and indicated for FGG procedure (28)
* Good systemic health with absence of active periodontal disease
* Plaque and bleeding index <20%

Exclusion Criteria:

* Uncontrolled systemic disease
* Heavy smokers (> 10 cigarettes per day)
* Restorations that cannot be removed for proper treatment
* Pregnant or lactant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Volumetric changes of keratinized tissue (KT) around teeth after free gingival graft (FGG). | 6 weeks, 3 months, 6 months, 1 year
  A digital scan of the arch will be performed with an optical 3D measurement system (3Shape Trios) creating STL files. The corresponding reference and follow-up examinations of each clinical case will be virtually overlaid and combined into a common coordinate system (Geomagic, 3D Systems) using the Control X tool. By using of the buccal surfaces of the affected teeth as reference points for the superposition of the different time points
Colorimetric changes of keratinized tissue (KT) around teeth after free gingival | 6 weeks, 3 months, 6 months, 1 year
  A spectrophotometer (Easy Shade, VITA) will be used for the evaluation of the gingiva color. Before each measurement, the camera will be calibrated. To objectively measure gingiva discoloration, spectrophotometric measurements of the buccal gingiva will be performed on the study and on the adjacent untreated control tooth. The spectrophotometer camera will be positioned perpendicular to the mid-buccal gum and two images will be captured at each site.The center of the area of interest will be located 1.5 mm apical to the mid-buccal gingival margin and 3 mm.
  The spectral analysis will generate the CIE-Lab (Commission Internationale d'Eclairage) color coordinates L: luminosity, a: chroma along the red-green axis and b: chroma along the yellow-blue axis. The total color difference DE between the gingiva will be calculated according to the formula DE = [(Limpl Lcontr) 2 + (aimpl acontr) 2 + (bimpl bcontr) 2] 1/2 (CIE 2004)

SECONDARY OUTCOMES:
Influence of the volume of an FGG on the color changes | 6 weeks, 3 months, 6 months, 1 year
  A spectrophotometer (Easy Shade, VITA) will be used for the evaluation of the gingiva color. Before each measurement, the camera will be calibrated. To objectively measure gingiva discoloration, spectrophotometric measurements of the buccal gingiva will be performed on the study and on the adjacent untreated control tooth. The spectrophotometer camera will be positioned perpendicular to the mid-buccal gum and two images will be captured at each site.The center of the area of interest will be located 1.5 mm apical to the mid-buccal gingival margin and 3 mm.
  The spectral analysis will generate the CIE-Lab (Commission Internationale d'Eclairage) color coordinates L: luminosity, a: chroma along the red-green axis and b: chroma along the yellow-blue axis. The total color difference DE between the gingiva will be calculated according to the formula DE = [(Limpl Lcontr) 2 + (aimpl acontr) 2 + (bimpl bcontr) 2] 1/2 (CIE 2004)
Influence of the volume of an FGG on the contraction of the keratinized gingiva | 6 weeks, 3 months, 6 months, 1 year
  Influence of the volume of an FGG on the contraction of the keratinized gingiva being evaluated with intraoral scans (IS) A digital scan of the arch will be performed with an optical 3D measurement system (3Shape Trios) creating STL files. The corresponding reference and follow-up examinations of each clinical case will be virtually overlaid and combined into a common coordinate system (Geomagic, 3D Systems) using the Control X tool. By using of the buccal surfaces of the affected teeth as reference points for the superposition of the different time points

CONTACTS AND LOCATIONS:
Locations (1):
- International University of Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided